CLINICAL TRIAL: NCT00848068
Title: Evaluation of FID 114657 on Tear Film Lipid Layer Thickness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C-07-61
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Dry Eye
Keywords: lipid layer thickness
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OD (Right Eye) (Other): FID 114657 or OPTIVE
  Interventions: Other: FID 114657; Other: OPTIVE Lubricant Eye Drops
- OS (Left eye) (Other): FID 114657 or OPTIVE
  Interventions: Other: FID 114657; Other: OPTIVE Lubricant Eye Drops

INTERVENTIONS:
Other: FID 114657 — artificial tears
Other: OPTIVE Lubricant Eye Drops — artificial tears

SUMMARY:
To evaluate the effects of FID 114657 on the tear film lipid layer thickness of patients with dry eye.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent document and HIPAA privacy document must be read, signed and dated by the patient or legally authorized representative before conducting any procedures.
* Patients (minimum age 18) with dry eye. Criteria for the diagnosis must include the following characteristics:

  * Positive response to the question, "Do you ever feel your eyes?";
  * Baseline LLT value of ≤75nm (OU), not varying by more than ±15 nm over the course of a 10-minute observation period, difference in LLT between the two eyes must be ≤15nm, and increase in LLT after three forceful blinks must be ≤15nm.
* Patients must have best-corrected Snellen visual acuity of 20/70 or better in each eye.
* Able and willing to follow study instructions.

Exclusion Criteria:

* Use of topical ocular drops within 12 hours of the study visit; or use of a topical ocular ointment within 36 hours of the study visit. In addition, use of any concomitant topical ocular drugs during the study period.
* History or evidence of ocular or intraocular surgery in either eye within the past six months.
* History or evidence of serious ocular trauma in either eye within the past six months.
* History of intolerance or hypersensitivity to any component of the study medications.
* History of and/or current evidence of glaucoma or ocular hypertension in either eye.
* History of and/or current evidence of active intraocular inflammation in either eye (i.e., retina/macula/choroid).
* History or evidence of epithelial herpes simplex keratitis (dendritic keratitis); vaccinia; active or recent varicella viral disease of the cornea and/or conjunctiva; ocular rosacea; chronic bacterial disease of the cornea and/or conjunctiva and/or eyelids; mycobacterial infection of the eye; and/or fungal disease of the eye.
* Ocular conditions such as active acute blepharitis, conjunctival infections, iritis, conjunctival abnormalities (including pinguecula greater than 1mm in diameter, located closer than 2mm to the limbus or elevated more than 0.2mm), eyelid abnormalities (including entropion and ectropion) or any other ocular condition that may, in the opinion of the investigator, preclude the safe administration of the test articles.
* Patients using systemic medications that may contribute to dry eye (e.g. cold and allergy medications, tricyclic antidepressants, hormone replacement therapies) may not be enrolled in the study unless they have been on a stable dosing regimen for a minimum of 30 days prior to the study visit.
* Any ocular or systemic medical condition that might influence the tear film (other than dry eye).
* Individuals unwilling to discontinue contact lens wear during the study period. Contact lens wear must have been discontinued a minimum of 12 hours prior to the study visit.
* Individuals unwilling to discontinue use of cosmetics (such as eyeliner, mascara or eye shadow) or facial creams on or around the eyelids on the day of the study.
* Participation in an investigational drug or device study within 30 days of entering this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
lipid layer thickness | Instill assigned test article to the right eye and begin timing the examination process. Measure lipid layer thickness at 1 minute, 5 minutes, 15 minutes and 60 minutes post instillation